CLINICAL TRIAL: NCT06948916
Title: Investigation of the Validity and Reliability of 6-minute Pegboard and Ring Test in Patients With Interstitial Lung Disease
Brief Title: Validity and Reliability of 6-minute Pegboard and Ring Test in Patients With Interstitial Lung Disease
Status: Recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: 2024 - 1688
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Interstitial Lung Diseases (ILD); Exercise Capacity; Upper Extremity
Keywords: Interstitial lung diseases; Exercise Capacity; Upper extremity
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ILD: Patients diagnosed with ILD according to ATS/ERS criteria

SUMMARY:
Interstitial lung diseases (ILD) are a heterogeneous group of chronic respiratory diseases that cause significant mortality and morbidity worldwide, characterized by diffuse inflammation in the lung parenchyma and vascular structures, can progress to fibrosis, have known or unknown etiology, and can develop secondary to systemic autoimmune connective tissue diseases other than diseases where the primary pathology is in the lung. The 6-minute peg-board and ring test, which was first developed to determine the upper extremity exercise capacity of chronic obstructive pulmonary disease patients, is an exercise test used to evaluate upper extremity functional exercise capacity in different lung diseases. It has been determined that there is no study on the validity and reliability of this test in individuals with ILD.

DETAILED DESCRIPTION:
Interstitial lung diseases (ILD) are chronic respiratory diseases that cause significant mortality and morbidity worldwide. The 6-minute peg-board and ring test, which was first developed to determine the upper extremity exercise capacity of chronic obstructive pulmonary disease patients, is an exercise test used to evaluate upper extremity functional exercise capacity in different lung diseases. It has been determined that there is no study on the validity and reliability of this test in individuals with ILD. In this patient group, the upper extremity muscles are seriously affected. In addition, serious desaturation develops during exercise tests that require walking and the use of larger muscle groups, such as the 6-minute walking test. For this reason, upper extremity aerobic exercise capacity gains importance in this patient group. There are no studies in the literature on the validity and reliability of 6-PBRT in patients with ILD, although its validity and reliability have been studied in different patient groups such as COPD, PAH, and asthma. The primary aim of our study was to determine the validity and reliability of the 6-minute peg-board and ring test for patients with interstitial lung disease.

The study will be conducted between June 2023 and February 2025 on patients diagnosed with interstitial lung disease who were referred to the Cardiopulmonary Rehabilitation Unit of the Department of Physiotherapy and Rehabilitation, Faculty of Medicine, Gazi University for rehabilitation by the Department of Chest Diseases, Faculty of Medicine, Gazi University. Data from patients who have been followed up will be analyzed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ILD according to ATS/ERS criteria,
* Ages between 18 and 75,
* Pulmonary infection during the previous month,
* Participants who voluntarily participated in the study were included.

Exclusion Criteria:

* Patients were excluded if they had:
* Acute pulmonary exacerbation or respiratory infection in the last four weeks
* Obstructive lung disease
* Systemic conditions affecting neurological, neuromuscular, orthopedic, or physical functions
* Recent participation in a planned exercise program (within three months)
* Cognitive impairment affecting exercise test understanding
* Contraindications to exercise testing per the American Sports Medicine Association
* Cancer, renal, or hepatic disease
* Aortic stenosis, complex arrhythmia, or aortic aneurysm
* Serious cardiovascular diseases like uncontrolled hypertension, diabetes, heart failure, or arrhythmia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female and Male
Study Population: Patients diagnosed with ILD
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-07-12 (Estimated); Study Completion 2025-08-12 (Estimated)

PRIMARY OUTCOMES:
Upper extremity functional exercise capacity | Trough study completion, an average of 1 year
  To evaluate upper extremity functional exercise capacity, 6-minute pegboard and ring tests will be applied twice with 15-30 minute intervals. Before the test, individuals will be seated and rested for at least 10 minutes. Individuals will be provided with detailed information about the application of the test before the test. Patients will be informed not to interfere with rings that fall during the test and to continue the test. It will be explained that they can stop and rest if they feel too uncomfortable to continue the test, but this time will be included in the test duration. Before the actual test, subjects will be allowed to move up and down one loop as a practice to learn the test procedure. As a test result, the total number of rings worn at the end of six minutes will be recorded in numbers.

SECONDARY OUTCOMES:
Upper Extremity Maximal Exercise Capacity | Trough study completion, an average of 1 year
  Upper extremity maximal exercise capacity will be assessed by symptom-limited cardiopulmonary exercise testing on arm ergometer at gradually increasing workload, and oxygen consumption will be measured during the test.
Upper extremity activities of daily living | Trough study completion, an average of 1 year
  Limitations in upper extremity activities of daily living will be assessed with the Milliken Activities of Daily Living Scale (ACS), a patient-reported outcome measure. The Turkish validity-reliability study was conducted by Semin Akel and colleagues in 2012. The scale contains 47 items related to different activities of daily living, including meal preparation, eating, personal care, self-dressing, handling objects, house cleaning, laundry, and other activities. There is an integrated scoring procedure that uses the multiplication of each ability score by each requirement score, yielding a possible score of 15 for each item and a possible total integrated score of 705. The total score was used in this study. Lower scores indicate greater limitations in the ability to perform daily tasks with the upper extremities.
Dyspnea | Trough study completion, an average of 1 year
  The assessment of dyspnea at rest, during, and after exercise training will be made with the Modified Borg scale. The Modified Borg scale is a subjective scale and scores the shortness of breath at rest and/or during activity between 0-10. The lowest score of 0 (zero) indicates 'none', and the highest score of 10 (ten) indicates 'maximal' shortness of breath. The Modified Medical Research Council (MMRC) dyspnea scale will be used to determine the perception of dyspnea during activities of daily living. The London Chest Activities of Daily Living Scale, developed by Garrod et al. to examine dyspnea that occurs with daily living activities in chronic obstructive pulmonary disease and whose Turkish validity and reliability were performed by Saka et al., will be used to assess shortness of breath that occurs during activities of daily living.
Respiratory Muscle Strength | Trough study completion, an average of 1 year
  Maximal inspiratory and expiratory muscle strength will be evaluated using mouth pressure device.
Peripheral muscle strength | Trough study completion, an average of 1 year
  Shoulder flexor and shoulder abductor muscle strength will be assessed with a portable handheld dynamometer (JTECH Power Track Commander, Baltimore, USA).
Disease Related Quality of life | Trough study completion, an average of 1 year
  The Saint George Respiratory Questionnaire is a questionnaire used to assess the quality of life in respiratory diseases and its Turkish validity and reliability were conducted by Polatlı et al. The questionnaire consists of 3 sections: symptoms (8 items), activities (16 items), and effects of the disease (26 items) and a total of 50 items: The 3 sections of the test are scored separately. Then, a total score is obtained. The total score varies between 0-100. A score of zero is normal, while a score of 100 indicates maximum disability. As the total score increases, it indicates that the patients' quality of life is poor.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | Trough study completion, an average of 1 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, forced expiratory volume in the first second (FEV1) will be evaluated.
Pulmonary function (Forced vital capacity (FVC)) | Trough study completion, an average of 2 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, forced vital capacity (FVC) will be evaluated.
Pulmonary function (FEV1/FVC) | Trough study completion, an average of 1 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, FEV1 / FVC will be evaluated.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | Trough study completion, an average of 1 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be evaluated.
Pulmonary function (Peak flow rate (PEF)) | Trough study completion, an average of 1 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, peak flow rate (PEF) will be evaluated.
Pulmonary function (Diffusion capacity for carbon monoxide (DLCO)) | Trough study completion, an average of 1 year
  Carbon monoxide diffusing capacity of the lung (DLCO) is a measurement to assess the lungs' ability to transfer gas from inspired air to the bloodstream. Its measurement uses carbon monoxide to calculate the pulmonary diffusion capacity. The most common method is the standard single-breathe diffusing capacity test. It is expressed in mmol/(min*kPa) and as a percentage (%) of the expected value.

CONTACTS AND LOCATIONS:
Overall Officials: Meral BOŞNAK GÜÇLÜ, Prof. Dr., Study Director — Gazi University; Nazire Nur YILDIZ, M.Sc., Study Chair — Nigde Omer Halisdemir University; Nilgün YILMAZ DEMİRCİ, Prof. Dr., Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
To protect patient data, it will not be shared.

REFERENCES:
- See also: Celli BR, Rassulo J, Make BJ. Dyssynchronous breathing during arm but not leg exercise in patients with chronic airflow obstruction. New England Journal of Medicine. 1986;314(23):1485-90. — https://pubmed.ncbi.nlm.nih.gov/3702963/
- See also: Zhan S, Cerny FJ, Gibbons WJ, Mador MJ, Wu Y-W. Development of an unsupported arm exercise test in patients with chronic obstructive pulmonary disease. Journal of Cardiopulmonary Rehabilitation and Prevention. 2006;26(3):180-7. — https://pubmed.ncbi.nlm.nih.gov/16738459/
- See also: Kahraman BÖ, Özsoy İ, Tanrıverdi A, Akdeniz B, Özpelit E, Şentürk B, et al. Validity and reliability of the 6-minute pegboard ring test in patients with pulmonary hypertension. Türk Fizyoterapi ve Rehabilitasyon Dergisi. 2020;31(2):210-7. — https://dergipark.org.tr/en/download/article-file/1036390
- See also: Calik-Kutukcu E, Tekerlek H, Bozdemir-Ozel C, Karaduz BN, Cakmak A, Inal-Ince D, et al. Validity and reliability of 6-minute pegboard and ring test in patients with asthma. Journal of Asthma. 2022;59(7):1387-95. — https://pubmed.ncbi.nlm.nih.gov/33985406/
- See also: Takeda K, Kawasaki Y, Yoshida K, Nishida Y, Harada T, Yamaguchi K, et al. The 6-minute pegboard and ring test is correlated with upper extremity activity of daily living in chronic obstructive pulmonary disease. International Journal of Chronic Obstructi — https://pubmed.ncbi.nlm.nih.gov/23901268/